CLINICAL TRIAL: NCT06341335
Title: A Randomized, Double-blind, Phase 3 Study Of Cadonilimab (AK104) Plus Pulocimab (AK109) And Paclitaxel Versus Paclitaxel In Patients With Advanced Gastric Or Gastroesophageal Junction Adenocarcinoma Who Failed First-line Immunochemotherapy
Brief Title: A Study of AK104/Placebo Plus AK109/Placebo And Paclitaxel in Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK109-301
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Gastric and Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cadonilimab in combination with pulocimab and paclitaxel (Experimental): Cadonilimab (AK104) in combination with pulocimab (AK109) and paclitaxel, iv, every 3 weeks
  Interventions: Drug: cadonilimab; Drug: pulocimab; Drug: paclitaxel
- Placebo in combination with paclitaxel (Active Comparator): Placebo in combination with Paclitaxel, iv, every 3 weeks
  Interventions: Drug: paclitaxel; Drug: placebo

INTERVENTIONS:
Drug: cadonilimab — iv, q3w
  Other Names: AK104
  Arms: Cadonilimab in combination with pulocimab and paclitaxel
Drug: pulocimab — iv, q3w
  Other Names: AK109
  Arms: Cadonilimab in combination with pulocimab and paclitaxel
Drug: paclitaxel — iv, q3w
Drug: placebo — iv, q3w
  Arms: Placebo in combination with paclitaxel

SUMMARY:
This randomized, multicenter, double-blind, phase 3 study will evaluate the efficacy and safety of the combination of cadonilimab (AK104) and pulocimab (AK109) and paclitaxel compared with paclitaxel in patients with advanced gastric or gastroesophageal junction adenocarcinoma who failed first-line immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 18 years and ≤ 75 years
3. Histologically or cytologically documented advanced unresectable or metastatic gastric adenocarcinoma or gastroesophageal Junction (GEJ) adenocarcinoma.
4. Failed first-line treatment with PD-(L)1 monoclonal antibody and standard chemotherapy
5. At least one measurable disease based on RECIST v1.1
6. ECOG status of 0 or 1
7. Estimated survival ≥ 3 months
8. Adequate organ function per protocol-defined criteria
9. Women of childbearing potential and men with female partners of childbearing potential must agree to use effective contraception during treatment and for at least 120 days following the last dose of study treatment

Exclusion Criteria:

1. Mixed gastric or gastroesophageal Junction cancer containing other pathological components than adenocarcinoma
2. HER2-positive
3. Known other invasive malignancies within 3 years
4. Subjects who are currently participating in other interventional study
5. Received prior systemic anti-tumour therapy within 4 weeks before randomization
6. Previous systemic treatment with taxane within 6 months before randomization
7. Previous systemic treatment targeting VEGF or anti-VEGFR signaling pathways
8. In addition to anti-PD-(L)1 monoclonal antibody, prior exposure to other immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy or other therapy that targets anti-tumor immune mechanisms
9. History of immune-related adverse effects leading to recommendation against reintroduction of immunotherapy or any condition dependency on systemic therapy with glucocorticoids or immunosuppressive agents within 14 days prior to randomization
10. History of severe infection within 4 weeks prior to randomization
11. Presence of central nervous system metastases, leptomeningeal metastases, or spinal cord compression
12. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage
13. History or presence of a serious hemorrhage or known bleeding tendency within 2 months before randomization
14. Major surgical procedure or serious trauma within 28 days prior to randomization
15. History of interstitial lung disease or noninfectious pneumonitis
16. Active infectious diseases, including tuberculosis, HIV infection, syphilis infection，or hepatitis B/C
17. Known allergy to the antibody or any component of the study drug; Or the constitution of being allergic to multiple substances
18. History of allogeneic organ transplantation or allogeneic haematopoietic stem cell transplantation
19. Toxicities of prior anticancer therapy have not resolved to ≤ Grade 1 (NCI-CTCAE version 5.0)
20. Use of live vaccines within 30 days prior to randomization
21. Pregnant or lactating women.
22. Any condition considered by the investigator to be inappropriate for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by blinded independent central review (BICR) | Up to 2 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first (based on RECIST 1.1 criteria).
Overall survival (OS) | Up to 2 years
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed by investigator | Up to 2 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first (based on RECIST 1.1 criteria).
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as proportion of subjects who have a complete or partial response relative to baseline according to RECIST 1.1 criteria
Duration of Response (DoR) | Up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression(based on RECIST v1.1 criteria) or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (based on RECIST v1.1 criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Xiaotian Zhang, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China